CLINICAL TRIAL: NCT06205368
Title: Evaluating the Effectiveness of a Mobile HIV Prevention Application to Increase HIV and STI Testing and PrEP Initiation Among Rural Men Who Have Sex With Men
Brief Title: Evaluating the Effectiveness of a Mobile HIV Prevention App to Increase HIV and Sexually Transmitted Infections (STI) Testing and PrEP Initiation Among Rural Men Who Have Sex With Men
Acronym: CombineApp
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jeb Jones, Professor, Emory University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00006280; R01MH134267-01 (NIH)
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: HIV Infections; STI; HIV Pre-exposure Prophylaxis
Keywords: GBMSM; PrEP; HIV; Gay; HIV prevention; STI testing; HIV testing
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases; Homosexuality | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Combine app with all features except the ability to order self-test kits (Other): Participants will receive a modified standard of care which consists of the Combine app with all features except the ability to order self-test kits. The HIV/STI testing locator in the app will be available.
  Interventions: Behavioral: Combine mobile app
- Combine app + motivational interview (Other): In addition to the other Combine app features, participants will receive a motivational interview within 4 weeks of downloading the app.
  Interventions: Behavioral: Combine mobile app; Behavioral: Motivational interview
- Combine app + ability to order up 2 free HIV/STI self-test kits (Other): In addition to the other Combine app features, participants in this arm will be able to order up to two HIV/STI self-test kits at no charge during each year of follow-up.
  Interventions: Behavioral: Combine mobile app; Behavioral: HIV/STI testing
- Combine app + motivational interview + ability to order HIV/STI test kits via the app (Other): In addition to the other Combine app features, participants in this arm will receive both the motivational interview and the ability to order HIV/STI test kits via the app.
  Interventions: Behavioral: Combine mobile app; Behavioral: Motivational interview; Behavioral: HIV/STI testing

INTERVENTIONS:
Behavioral: Combine mobile app — * HIV/STI testing: learn more about testing options; create a plan to test 1-4 times in the coming year; locate places for those tests and/or order at-home test kits; and schedule reminders for periodic testing
  * Pre-exposure prophylaxis: PrEP self-assessment at first app use; monthly rescreening for PrEP eligibility; recommendation for PrEP based on Centers for Disease Control and Prevention (CDC) criteria; PrEP provider locator.
  * Behavioral risk assessment: e.g. HIV risk behaviors; sex while drunk or high, condomless anal intercourse with a positive or unknown HIV status partner, multiple sex partners, recent STI diagnosis, use of drugs) and protective behaviors
  * Non-occupational post-exposure prophylaxis (nPEP): information about nPEP; self-assessment; locator; referral to PrEP for men who evaluate multiple exposures for nPEP indication
  * Product ordering: participants can order condoms, condom-compatible lubricants, and at-home STI specimen collection kits.
  Other Names: Mobile app
Behavioral: Motivational interview — The interview will be grounded in the Social Cognitive Theory of self-regulation (SCT) to reflect the underlying theory of the Combine app. It will be designed to enhance the effectiveness of the app by highlighting app features (e.g., frequently asked questions, product ordering, testing locators) and discussing strategies for following through on goals related to sexual health (e.g., creating and adhering to a testing plan)
  Arms: Combine app + motivational interview; Combine app + motivational interview + ability to order HIV/STI test kits via the app
Behavioral: HIV/STI testing — Participants will be able to order free HIV/STI self-test kits; they will be able to order up to two sets of kits during each of years 1 and 2 of follow-up. HIV and STI test kit orders are independent: ordering an HIV test kit does not trigger shipment of an STI kit and vice versa. When an order is placed, kits containing biospecimen self-collection tools are shipped directly to the participant along with written instructions and a link to video instructions on how to collect each of the samples (e.g., urine, rectal, blood). Return packaging is enclosed with instructions for participants to locate a drop-off location to return their samples to the lab.
  Arms: Combine app + ability to order up 2 free HIV/STI self-test kits; Combine app + motivational interview + ability to order HIV/STI test kits via the app

SUMMARY:
The goal of this clinical trial is to test the efficacy of a mobile app, Combine, to increase the uptake of HIV and STI testing and pre-exposure prophylaxis (PrEP) over 24 months and to assess the effects of different implementation strategies on intervention maintenance among GBMSM in rural southern United States. The main aims of the study are:

* To assess the relative effects of three treatment conditions on gains in engagement in HIV prevention compared to a modified standard of care control condition
* Measure and assess secondary factors affecting app implementation
* Refine implementation strategies and coordinate with potential funders Participants will download an HIV prevention smartphone app and be randomly assigned to one of four groups:
* Control: App access only
* Self-testing: App access + ability to order HIV and STI self-test kits
* Motivational interview: App access + motivational interview to develop plans to use app effectively.
* Self-testing + motivational interview: App access + ability to order HIV and STI self-test kits + motivational interview to develop plans to use app effectively.

Researchers will compare each of the latter three groups to the control condition to see if HIV and STI testing increase in these groups

DETAILED DESCRIPTION:
The uptake of HIV and STI testing among gay and bisexual men who have sex with men (GBMSM) in the rural southern US is low. However, HIV and STI testing is a fundamental gateway to preventive services, such as PrEP, and treatment provision. Thus, the research team must identify methods to increase the uptake of HIV and STI testing among this population that experiences disproportionate HIV and STI incidence. The research team has developed an app, Combine, that is an adaptation of HealthMindr, an app that has demonstrated efficacy in increasing the uptake of HIV testing among urban GBMSM. Combine was adapted using input from GBMSM in rural areas to address issues specific to this population such as increased experiences of stigma and reduced access to culturally competent care. The investigator proposes to conduct a Type 2 Hybrid Effectiveness-Implementation randomized controlled trial to test the efficacy of Combine to increase uptake of HIV and STI testing over 24 months of follow-up and to examine the effect of different implementation strategies among GBMSM in the rural South. Combine will include components for self-administered risk assessments, developing and supporting a plan for frequent HIV and STI testing, information about PrEP, and PrEP and HIV/STI testing provider locators. Previous trials of app-based HIV prevention have included the ability to order free HIV and STI self-test kits. However, there is no consensus among health officials around whether at-home self-tests are an optimal solution for increasing HIV and STI testing. Additionally, despite the availability of free HIV and STI self-test kits in previous studies, large proportions of men still do not complete HIV tests, and even fewer complete STI tests. Thus, the investigator will evaluate the effect of two different intervention components on HIV and STI uptake in a 2x2 factorial trial design: availability of HIV and STI self-test kits ordered through the app and a motivational interview designed to enhance the existing app content, increased self-efficacy to develop and follow through with a testing plan, and develop strategies to deal with experiences of stigma.

The investigator will assess the main effects of the availability of HIV and STI self-test kits and the motivational interview on HIV and STI testing uptake, PrEP initiation, and intervention maintenance over 24 months of follow-up. The investigator's community-based partner, Engaging Arkansas Communities, will work with the research team through all stages of the project to ensure that the team is obtaining the necessary data to inform future implementation.

ELIGIBILITY:
Inclusion criteria

* Assigned male at birth and currently identifies as male
* Age 18-45 years, inclusive
* Reside in the U.S. South as defined by the Census Bureau or in Missouri
* Reside in a county classified as rural using the Index of Relative Rurality
* Have an Android or iPhone operating system (iOS) phone with active service
* Willing to download a study app to their phone
* English speaker
* Report anal sex with a man in the past 12 months
* HIV-negative or unknown serostatus
* Not currently using PrEP

Exclusion criteria

- Unable to provide consent

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Assigned male at birth and currently identifies as male
Enrollment: 473 (Actual)
Dates: Start 2024-03-27 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Uptake of HIV testing | Screening, Month 6, Month 12, Month 18, Month 24
  The investigator will look at the change in number of participants getting tested for HIV by using online surveys. Uptake of testing will be defined as ordering, using, and returning a kit for laboratory analysis or obtaining a test at an in-person provider and reporting the result.
Uptake of STI testing | Screening, Month 6, Month 12, Month 18, Month 24
  The investigator will look at the change in number of participants getting tested for STIs by using online surveys. Uptake of testing will be defined as ordering, using, and returning a kit for laboratory analysis or obtaining a test at an in-person provider and reporting the result.
PrEP initiation | Screening, Month 6, Month 12, Month 18, Month 24
  The investigator will look at the change in number of participants taking PrEP over the course of the study. PrEP initiation will be defined as obtaining a new PrEP prescription for the first time or after a period of non-use of at least three months

CONTACTS AND LOCATIONS:
Overall Officials: Jeb Jones, PhD, Principal Investigator — Rollins School of Public Health
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Demographics and Primary Outcomes data will be shared upon request.
Supporting Information: Study Protocol, SAP
Time Frame: After the publication of primary outcome data
Access Criteria: Analyses that don't overlap with specific aims, per PI approval will be shared with those who request them from the PI via email.

REFERENCES:
- [Derived] Jones J, Manley G, Glynn TR, Wall KM, Baral SD, Harris ED, Benkeser D, Sullivan PS. Evaluating the Effectiveness of a Mobile HIV Prevention App to Increase HIV and Sexually Transmitted Infection Testing and Pre-Exposure Prophylaxis Initiation Among Rural Men Who Have Sex With Men in the Southern United States: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Jul 23;14:e69540. doi: 10.2196/69540. PMID 40699887

DOCUMENTS (1):
  • Informed Consent Form (2025-07-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT06205368/ICF_000.pdf